CLINICAL TRIAL: NCT03082235
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E6742 in Healthy Adult Subjects
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E6742 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: E6742-A001-001
Record Dates: First submitted 2017-03-14; First posted 2017-03-17 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2017-11

CONDITIONS: Healthy Participants
Keywords: Healthy participants; E6742; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Cohort 1: 10 mg E6742 (Experimental): Participants will receive 10 milligrams (mg) E6742 as a single oral dose in the fasted state.
  Interventions: Drug: E6742
- Cohort 1: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state.
  Interventions: Drug: Placebo
- Cohort 2: 25 mg E6742 (Experimental): Participants will receive 25 mg E6742 as a single oral dose in the fasted state.
  Interventions: Drug: E6742
- Cohort 2: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state.
  Interventions: Drug: Placebo
- Cohort 3: 50 mg E6742 (Experimental): Participants will receive 50 mg E6742 as a single oral dose in the fasted state.
  Interventions: Drug: E6742
- Cohort 3: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state.
  Interventions: Drug: Placebo
- Cohort 4: 100 mg E6742 (Experimental): Participants will receive 100 mg E6742 as a single oral dose in the fasted state. Participants will then receive the same single oral dose of E6742 again in the fed state after a washout interval (at least 7 days or 5 half-lives of E6742, whichever is longer) for the evaluation of food effect.
  Interventions: Drug: E6742
- Cohort 4: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state. Participants will then receive the same single oral dose of placebo again in the fed state after a washout interval (at least 7 days ) for the evaluation of food effect.
  Interventions: Drug: Placebo
- Cohort 5: 200 mg E6742 (Experimental): Participants will receive 200 mg E6742 as a single oral dose in the fasted state.
  Interventions: Drug: E6742
- Cohort 5: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state.
  Interventions: Drug: Placebo
- Cohort 6: 400 mg E6742 (Experimental): Participants will receive 400 mg E6742 as a single oral dose in the fasted state.
  Interventions: Drug: E6742
- Cohort 6: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state.
  Interventions: Drug: Placebo
- Cohort 7: 800 mg E6742 (Experimental): Participants will receive 800 mg E6742 as a single oral dose in the fasted state.
  Interventions: Drug: E6742
- Cohort 7: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching E6742 in the fasted state.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6742 — gelatin capsules
  Arms: Cohort 1: 10 mg E6742; Cohort 2: 25 mg E6742; Cohort 3: 50 mg E6742; Cohort 4: 100 mg E6742; Cohort 5: 200 mg E6742; Cohort 6: 400 mg E6742; Cohort 7: 800 mg E6742
Drug: Placebo — gelatin capsules
  Arms: Cohort 1: Matching placebo; Cohort 2: Matching placebo; Cohort 3: Matching placebo; Cohort 4: Matching placebo; Cohort 5: Matching placebo; Cohort 6: Matching placebo; Cohort 7: Matching placebo

SUMMARY:
Study E6742-A001-001 is a randomized, double-blind, placebo-controlled, single ascending dose study conducted to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending oral doses of E6742 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking, male or female, age ≥18 years and ≤45 years old at the time of informed consent
* Body mass index (BMI) ≥18 and <32 kilograms per meters squared (kg/m2) at Screening

Exclusion Criteria:

* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 International Units per Liter [IU/L] or equivalent units of β-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation). No sperm donation is allowed during the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation.
* Any history of gastrointestinal surgery that may affect pharmacokinetic (PK) profiles of E6742 (eg, hepatectomy, nephrectomy, digestive organ resection) at Screening
* A prolonged QTcF interval (QTcF >450 ms) demonstrated on ECG at Screening or Baseline
* Persistent systolic blood pressure >130 mmHg or diastolic blood pressure >85 mmHg diastolic at Screening or Baseline Heart rate less than 50 or more than 100 beats/min at Screening or Baseline
* Known history of prolonged QT/QTc interval
* Left bundle branch block
* Known history of myocardial infarction or active ischemic heart disease
* Known history of clinically significant arrhythmia or uncontrolled arrhythmia
* Known history of clinically significant drug allergy at Screening
* Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening
* Known to be human immunodeficiency virus (HIV) positive at Screening
* Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse within the 2 years prior to Screening, or those who have a positive urine drug and alcohol test at Screening or Baseline
* Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
* Use of prescription drugs within 4 weeks before dosing
* Intake of over-the-counter (OTC) medications within 2 weeks before dosing
* Currently enrolled in another clinical study or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) before informed consent
* Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week before dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with any serious adverse event and number of participants with any non-serious adverse event | from Screening up to Day 7
  The number of participants with any serious adverse event and the number of participants with any non-serious adverse event will be reported.
Mean maximum observed concentration (Cmax) of E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Time at which the highest drug concentration occurs (tmax) for E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Area under the concentration-time curve from zero time to 24 hours postdose (AUC[0-24h]) E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Area under the concentration-time curve from zero time to 72 hours postdose (AUC[0-72h]) for E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC[0-t]) for E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Area under the concentration-time curve from zero time extrapolated to infinite time (AUC[0-inf]) for E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Terminal elimination phase half-life (t1/2) for E6742 and the metabolite ER-1132963 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Apparent total clearance following extravascular administration (CL/F) for E6742 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Apparent volume of distribution at terminal phase (Vz/F) for E6742 in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
AUC metabolite to E6742 ratio following molecular weight correction to E6742 equivalents in plasma | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose). Cohort 4: In both periods (Treatment Periods 1 [7 days] and 2 [6 days]), Day 1 at predose and 0.5 (30 minutes), 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose; Day 2 (24 and 36 hours postdose); Day 3 (48 hours postdose); Day 4 (72 hours postdose); Day 5 (96 hours postdose); Day 6 (120 hours postdose); Day 7 (144 hours postdose).
Amount of unchanged drug excreted in urine (Ae) for E6742 and the metabolite ER-1132963 | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Days 1 to 7: predose and 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose. Cohort 4: Days 1 to 7 (Treatment Period 1): predose and 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose.
Renal clearance (CLR) | Days 1 to 7
  Cohorts 1, 2, 3, 5, and 6: Days 1 to 7: predose and 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose. Cohort 4: Days 1 to 7 (Treatment Period 1): predose and 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose.

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No